CLINICAL TRIAL: NCT07386951
Title: Heart Rate Variability Biofeedback in Distress Regulation and Burnout Prevention Among Security Forces
Brief Title: Heart Rate Variability Biofeedback in Security Forces
Acronym: GNR-HRVB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PT-214/25
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Psychological Distress; Well-Being, Psychological; Burnout
Keywords: Heart rate variability biofeedback; HRV biofeedback; Burnout; Stress management; Psychological distress; Mental health promotion; Workplace well-being
MeSH Terms: conditions — Psychological Well-Being; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: A randomized, parallel-group clinical trial in which participants are allocated to either a 4-week heart rate variability biofeedback (HRV-BFB) training program or to a no-intervention control condition, with assessments at baseline, post-intervention (4 weeks), and 10-week follow-up.
Masking Description: Due to the nature of the intervention, participants and investigators are aware of who receive HRV biofeedback training or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRV Biofeedback Training (Experimental): Participants receive 12 individual sessions of heart rate variability biofeedback (HRV-BFB) over 4 weeks (one 12-minute session every 2 days). Training is delivered using a chest-worn ECG sensor (eSense Pulse) connected to a mobile application that provides real-time visual feedback.
  Interventions: Behavioral: Heart Rate Variability Biofeedback (HRV-BFB) Training
- Control: No Intervention (No Intervention): Participants receive no active intervention during the 4-week study intervention period and continue their usual duties and routines. They complete the same assessment schedule as the experimental group at baseline, 4 weeks, and 10 weeks. After completion of the final follow-up assessment, they are offered the opportunity to receive the HRV biofeedback training protocol.

INTERVENTIONS:
Behavioral: Heart Rate Variability Biofeedback (HRV-BFB) Training — Participants receive a structured heart rate variability biofeedback (HRV-BFB) training protocol delivered over 4 weeks. The intervention uses a portable chest-worn ECG sensor (eSense Pulse) connected via Bluetooth to a mobile application that provides real-time visual feedback of heart rate variability. Each participant completes 12 individual sessions of 12 minutes each (one session every 2 days). Sessions take place in a quiet room and follow a standardized format: a brief preparation phase, followed by approximately 10 minutes of guided breathing at resonance frequency (around 6 breaths per minute) using a visual breathing guide. The application displays color-coded feedback indicating how closely the participant's physiological response matches the target HRV pattern, and participants are instructed to adjust their breathing and recall positive memories to maximize time in the desired state. The aim is to increase HRV, strengthen parasympathetic activation, and improve stress and
  Other Names: HRV biofeedback; Resonance frequency breathing training
  Arms: HRV Biofeedback Training

SUMMARY:
This exploratory study evaluates the effectiveness of a 12-session Heart Rate Variability Biofeedback (HRV-BFB) protocol in reducing distress and burnout while promoting psychological well-being among Portuguese National Republican Guard (GNR) professionals. Exposed to high occupational stress from unpredictable risks, shift work, and limited resources, these individuals face elevated vulnerability to chronic stress outcomes. The intervention leverages real-time HRV feedback to enhance autonomic regulation, breathing techniques, and emotional self-regulation.

DETAILED DESCRIPTION:
Security forces like the GNR play a critical role in public safety but endure chronic stress from violence exposure, rapid decisions, shift rotations, and institutional resource shortages, heightening risks of distress, burnout, and impaired well-being. Distress arises when perceived threats exceed coping resources, leading to persistent negative emotions and health disruptions. Burnout manifests as exhaustion, mental distancing, and reduced efficacy from unmanaged chronic stress, with organizational impacts including absenteeism and eroded public trust. Psychological well-being encompasses multidimensional aspects like autonomy, relationships, and purpose beyond mere absence of illness. Traditional interventions face barriers such as stigma and access issues in rural GNR contexts, necessitating flexible, self-administered tools.

Intervention: HRV-BFB Protocol HRV-BFB trains participants to consciously modulate physiological responses via real-time monitoring of heart rate variability (HRV), reflecting sympathetic-parasympathetic balance. Low HRV links to mental health risks, while training targets resonance frequency breathing (~6 breaths/min or 0.1 Hz) to boost HRV amplitude, cardiac coherence, and baroreflex strength. Delivered autonomously via app post-initial guidance, the 12-session protocol requires no daily clinician oversight, enhancing accessibility for dispersed GNR personnel. Evidence shows HRV-BFB reduces stress, anxiety, depression, and burnout while fostering well-being in high-stress groups like emergency workers.

Study Objectives This exploratory trial tests whether HRV-BFB significantly lowers distress (multidimensional: physical, cognitive, emotional, behavioral), burnout levels, and boosts psychological well-being in GNR professionals. It aims to inform scalable interventions tailored to Portuguese police realities, addressing gaps in institutional support.

ELIGIBILITY:
Inclusion Criteria:

1. Operational military personnel of the Guarda Nacional Republicana (GNR) performing security, patrol, criminal investigation, or road safety duties
2. Any military rank or professional category within operational roles
3. Age between 18 and 55 years, inclusive
4. Both males and females
5. Capable of providing informed consent in Portuguese language

Exclusion Criteria:

1. Extended sick leave or medical absence
2. Currently involved in serious disciplinary proceedings
3. Use, modification, or initiation of psychotropic medication (including antidepressants, anti-anxiety medications, antipsychotics, mood stabilizers) within the past 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Psychological Distress (Kessler Psychological Distress Scale - K10) | Baseline (Week 0), Post-intervention (Week 4), Follow-up (Week 10)
  The Kessler Psychological Distress Scale (K-10) is a 10-item self-report measure assessing psychological distress over the past 30 days. Items measure anxiety and depressive symptoms on a 5-point Likert scale (1=never to 5=always). Total score range: 10-50 (higher scores indicate greater distress). Portuguese validation: α=0.91. Primary outcome is change from baseline to post-intervention (week 4) and follow-up (week 10).
Change in Occupational Burnout (Burnout Assessment Tool - BAT-12) | Baseline (Week 0), Post-intervention (Week 4), Follow-up (Week 10)
  The Burnout Assessment Tool Short Form (BAT-12) is a 12-item self-report measure of occupational burnout across 4 dimensions: exhaustion (3 items), mental distance (3 items), cognitive impairment (3 items), emotional impairment (3 items). 5-point Likert scale (1=never to 5=always). Total score range: 12-60. Portuguese validation: α=0.85. Primary outcome is change from baseline to post-intervention and follow-up.
Change in Psychological Well-Being (WHO-5 Well-Being Index) | Baseline (Week 0), Post-intervention (Week 4), Follow-up (Week 10)
  The WHO-5 Well-Being Index is a 5-item self-report measure of psychological well-being over the past 2 weeks. Items assess positive mood, vitality, sleep, daily functioning, and life satisfaction on a 0-5 scale. Total score range: 0-25 (higher=higher well-being). Primary outcome is change from baseline to post-intervention and follow-up.

SECONDARY OUTCOMES:
SDNN (Standard Deviation of NN Intervals) - Heart Rate Variability | Baseline (Week 0), after each of 12 training sessions
  SDNN measures the standard deviation of the average NN (R-R) intervals in milliseconds during a recording period. It is a general indicator of overall heart rate variability and reflects the body's overall capacity for physiological adaptation and autonomic flexibility. Higher SDNN values indicate better autonomic regulation.
RMSSD (Root Mean Square of Successive Differences) - Parasympathetic Activity | Baseline (Week 0), after each of 12 training sessions
  RMSSD measures the root mean square of successive differences between adjacent NN (R-R) intervals in milliseconds. It is a primary time-domain measure of high-frequency heart rate variability and specifically reflects parasympathetic (vagal) nervous system activity and the body's recovery capacity. Higher RMSSD indicates stronger parasympathetic tone.
Stress Index - Autonomic Balance Indicator | Baseline (Week 0), after each of 12 training sessions
  The Stress Index is a proprietary metric derived from heart rate variability analysis that quantifies autonomic nervous system balance. Lower values indicate better autonomic regulation and lower physiological stress levels. Higher values reflect sympathetic dominance and poorer stress adaptation.

CONTACTS AND LOCATIONS:
Locations (1):
- GNR - Comando Terrritorial de Setúbal (GNR - Setubal Territorial Command Centre), Setúbal, Portugal

IPD SHARING:
Plan to Share IPD: Undecided